CLINICAL TRIAL: NCT03082443
Title: The Effectiveness of a Group Intervention in the Nutritional Profile, Stress and Quality of Life in Patients in Cardiopulmonary Rehabilitation: a Randomized Clinical Trial
Brief Title: Group Intervention in the Nutritional Profile, Stress and Quality of Life in Patients in Cardiopulmonary Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Giana Freitas, Nutritionist, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 5287/16
Record Dates: First submitted 2017-02-16; First posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Stress; Quality of Life; Nutritional Status
Keywords: Cardiac rehabilitation; psychology; nutrition; stress; quality of life
MeSH Terms: interventions — Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic group (Experimental)
  Interventions: Other: Therapeutic group
- Control group (No Intervention)

INTERVENTIONS:
Other: Therapeutic group — The group will take place in six meetings lasting one hour. At the end of the intervention, a new group will be started.
  Issues related to illness, cardiopulmonary rehabilitation, aroused feelings and aspects of food education will be addressed, with the objective of improving nutritional profile, quality of life and reduction of stress level. During the meeting they will be constantly encouraged to express their feelings, doubts and exchanges of experiences.
  In the first individual care (both groups) an initial consultation will be performed when the sociodemographic and anthropometric data will be collected and the instruments will be applied: Lipp Adult Stress Inventory, SF-12 Quality of Life Assessment Questionnaire and Questionnaire Of Food Frequency. After three months, all participants will be reassessed by the psychologist and nutritionist and anthropometric data will be collected and the instruments applied again.
  Arms: Therapeutic group

SUMMARY:
To evaluate the effectiveness of a group intervention in the nutritional profile, in the stress and in the quality of life of patients in cardiopulmonary rehabilitation. Method: Randomized clinical trial using a semi-structured interview, sociodemographic and anthropometric data collection, with 164 participants divided into a control group and intervention group, the Food Frequency Questionnaire, the Lipp Adult Stress Symptom Inventory (ISSL) ) And the SF-12 Quality of Life Assessment Questionnaire. To verify the difference in nutritional profile, stress levels and quality of life between the groups, the chi-square test will be used for categorical variables and within each group the comparison between the moments will be through the MC Nemar test. In the quantitative variables the evaluation of the interaction between group and time will be through Variance Analysis using the design in Repeated Measures. Considering a significance level p <0.05. Expected Results: It is believed that psychological and nutritional intervention in patients participating in therapeutic groups helps them to elaborate questions regarding the difficulties of coping with the disease in the daily routine and to understand the importance of lifestyle care and healthy habits.

ELIGIBILITY:
Inclusion Criteria:

* Cardiopathy patients over 18 years of age, users of the Center for Cardiopulmonary and Metabolic Rehabilitation of the Cardiology Institute who signed the Term of Free and Informed Consent

Exclusion Criteria:

* Patients not able to respond to questionnaires at the time of application. Patients who do not want to continue responding to the survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2017-04-01 (Estimated); Primary Completion 2017-06 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants in a therapeutic group of patients in cardiac rehabilitation evaluated for stress | Six weeks
  For the evaluation of the patients will be used semi-structured interview, sociodemographic data, with 164 participants divided into a control group and intervention group, the Lipp Adult Stress Symptom Inventory (ISSL) will be applied.
Number of participants in a therapeutic group of patients in cardiac rehabilitation evaluated for quality of life | Six weeks
  For the evaluation of the patients will be used semi-structured interview, sociodemographic data, with 164 participants divided into a control group and intervention group,the SF-12 Quality of Life Assessment Questionnaire will be applied.
Number of participants in a therapeutic group of patients in cardiac rehabilitation evaluated for nutritional profile | Six weeks
  For the evaluation of the patients will be used semi-structured interview, sociodemographic and anthropometric data (weight, height, body mass index and waist circumference), with 164 participants divided into a control group and intervention group, The Food Frequency Questionnaire will be applied.